CLINICAL TRIAL: NCT01865825
Title: PPI Responsive Esophageal Eosinophilia: GERD or Eosinophilic Esophagitis?
Brief Title: Proton Pump Inhibitor (PPI) Responsive Eosinophilic Esophagitis EoE: Gastroesophageal Reflux Disease (GERD) or Eosinophilic Esophagitis (EoE)?
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jeffrey A Alexander, Principal Investigator, Mayo Clinic
Other Study IDs: 12-009305
Record Dates: First submitted 2013-05-23; First posted 2013-05-31 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Erosive Esophagitis
Keywords: Erosive Esophagitis; Gastroesophageal reflux disease
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Esophageal barium xray: We will recruit 20 patients with GERD without dysphagia for an esophageal barium xray for esophageal diameter measurements.
  The 20 Gastroesophageal Reflux Disease (GERD) patients will complete the Mayo Dysphagia Questionnaire 30-day and the Eosinophilic Esophagitis Actitivy Index (EEsAI) questionnaires
  Interventions: Radiation: Esophageal Barium Xray

INTERVENTIONS:
Radiation: Esophageal Barium Xray — •Fast for 4 hours prior to the Esophagram (upper GI x-ray). You will drink a liquid that has barium or another contrast agent in it. The radiologist will use the X-ray machine to look at your upper GI tract while you drink the contrast liquid. The x-ray exam should take between 10-15 minutes.
  We will have patients complete the Mayo Dysphasia Questionnaire-30 day.
  Other Names: GERD; Erosive Esophagitis

SUMMARY:
The investigators would like to determine if there are patients with PPI responsive Eosinophilic Esophagitis Infiltration that have significant loss of esophageal distensibility suggestive of esophageal fibrosis typical of classic Eosniophilic Esophagitis.

If this group of patients exists, the investigators would like to determine if they have the typical endoscopic features of EoE rather than those of GERD.

ELIGIBILITY:
Inclusion criteria:

* Age 18 or older
* Have either mild-to-moderate Los Angeles (LA) Classification System grade B, moderately severe LA grade C, or severe LA grade D erosive reflux esophagitis
* Or patients having a clinically indicated pH/impedance monitoring on proton pump inhibitor therapy for indications of gastroesophageal reflux disease.

Exclusion criteria:

* Neoplasm of the esophagus or stomach
* Inability to read due to: Blindness, cognitive dysfunction, or English language illiteracy
* Disorders which predispose to unreliable responses such as Schizophrenia, Alzheimer's disease or significant memory loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with GERD that have been currently diagnosed with erosive esophagitis at endoscopy, at Mayo Clinic Rochester, Minnesota
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Abnormal esophageal distensibility in patients with PPI responsive Eosinophilic Infiltrates to patients with Eosionophilic esophagitis and Gastroesophageal Reflux Disease. | 1 year
  We will evaluate endoscopic features of Gastroesophageal Reflux Disease(GERD) by reviewing endoscopic reports and images. The presence of esophageal narrowing, furrows, rings, fragility, and white spots will be noted form the endoscopic reports prior to the initiation of the Provation report system. We will review the endoscopic reports and the endoscopic photographs on those patients evaluated after the Provation report system was initiated. All images will be reviewed by one investigator unaware of the subjects clinical data and name

SECONDARY OUTCOMES:
The relationship of abnormal esophageal distensibility to other endoscopic findings of EoE (furrows, rings, fragility, stricture) | 1 year
  After reviewing endoscopic features of GERD by reviewing endoscopic reports and images. The presence of esophageal narrowing, furrows, rings, fragility, and white spots will be noted form the endoscopic reports prior to the initiation of the Provation report system. We will determine the relationship of abnormal esophagus distensibility to the endoscopic findings

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Alexander, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States